CLINICAL TRIAL: NCT01375153
Title: Effects of Brain Natriuretic Peptide on Appetite-regulating Hormones and Endothelial-derived Peptides
Brief Title: Brain Natriuretic Peptide Effects on Appetite Regulating Hormones and Endothelial Derived Peptides
Acronym: BNP/Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Anton Luger, Professor, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 060/2009
Record Dates: First submitted 2011-05-31; First posted 2011-06-17 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: BNP administration; appetite; ghrelin; PYY
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0,9% NaCl administered as a continuous intravenous infusion during four hours.
  Interventions: Drug: 0.9% NaCl
- BNP (Active Comparator): 3.0 pmol/kg/min human active BNP administered as a continuous intravenous infusion during four hours.
  Interventions: Drug: BNP

INTERVENTIONS:
Drug: BNP — 3.0 pmol/kg/min human active BNP administered as a continuous intravenous infusion during four hours
  Arms: BNP
Drug: 0.9% NaCl — 0.9% NaCl administered as a continuous intravenous infusion during four hours
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
Chronic heart failure is accompanied by anorexia and increased release of B-type natriuretic peptide (BNP) from the ventricular myocytes. The pathophysiological mechanisms linking heart failure and appetite-regulation remain unknown. This study aims to examine the impact of exogenous BNP administration on subjective ratings of hunger and satiety, and on appetite-regulating hormones in a placebo-controlled cross-over study performed in ten healthy human volunteers.

DETAILED DESCRIPTION:
This is a prospective, single blinded randomized, placebo-controlled, cross-over study, which will be conducted in ten healthy volunteers.

Each subject will participate in two study days/sessions, separated by a washout period of at least two weeks. The sessions will last approximately 4.5 hours. The subjects will come after having fasted overnight. Two intravenous cannulas will be placed in the right and left antecubital vein for infusions and blood sampling, respectively.

The subjects will receive intravenously once placebo and once 3.0 pmol/kg/min human active BNP (BNP-32) as a continuous intravenous infusion given during 4 hours (between time points 0 and 240 minutes). The order of study drugs will be randomized.

During the whole study session (lasting about 4.5 hours) the subject will remain fasted and confined to bed rest.

The changes in subjective ratings of hunger and satiety over time will be evaluated by 100 mm visual analog scales (VAS) half-hourly (between time points 0 and 240 minutes). Herewith the subjects rate their feeling of hunger (Hunger-VAS forms include the question: How hungry do you feel? Subjects are required to mark their feeling of hunger in a scale from 0 to 100 mm) and satiety (Satiety-VAS forms include the question: How satt do you feel? Subjects are required to mark their feeling of hunger in a scale from 0 to 100 mm).

Blood samples will be withdrawn twice at baseline (time points -5 minutes and 0 minutes) and hourly afterwards. Samples will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C for the later measurement of ghrelin, peptide YY, adiponectin, corticotropin, cortisol, adrenaline, noradrenaline, insulin, adrenomedullin, endothelin, copeptin, growth differentiation factor 15, BNP and atrial natriuretic peptide. All assays will be performed using commercial radioimmunoassays and enzyme-linked immunosorbent assays at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.

The changes in VAS and hormone concentrations over time will be evaluated using repeated measurements analysis of variance (ANOVA) using the SPSS release 12.0.1 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 40 years
* written informed consent
* BMI < 25 kg/m2
* no concomitant diseases
* BNP level within the normal range
* Normal renal function (serum creatinine of less then 1.2 mg/dL and/or creatinin clearance greater than 80ml/min)

Exclusion Criteria:

* systolic blood pressure < 90 mmHg
* impaired glucose tolerance or diabetes mellitus
* hyperthyroidism, hypothyroidism
* hepatic, renal or cardiovascular diseases
* malignancies
* history of medical therapy within 3 weeks prior to enrolment into the study
* history of anaphylaxis

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Changes in hunger scores on the visual analog scales (VAS) over time as compared to baseline (measured in mm) | Time points -5, 0, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
  Subjects will be asked to rate their feeling of hunger in 100 mm VAS half-hourly (between time points 0 and 240 minutes).
  Hunger-VAS forms include the question: How hungry do you feel? Subjects are required to mark their feeling of hunger in a scale of 0 to 100 mm.
Changes in satiety scores on the VAS over time as compared to baseline (measured in mm) | Time points -5, 0, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
  Subjects will be asked to rate their feeling of satiety in 100 mm VAS half-hourly (between time points 0 and 240 minutes).
  Satiety-VAS forms include the question: How satt do you feel? Subjects are required to mark their feeling of satiety in a scale of 0 to 100 mm.
Changes in plasma concentrations of ghrelin and acylated ghrelin over time as compared to baseline | Timepoints -5, 0, 60, 120, 180 and 240 minutes.
  Blood samples will be withdrawn from an intravenous cannula placed circa 10 minutes before the start of the study in the left antecubital vein. Samples will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C for the later measurement of ghrelin and acylated ghrelin. All assays will be performed using commercial assay kits at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.
Changes in plasma concentrations of peptide YY (PYY) over time as compared to baseline | Timepoints -5, 0, 60, 120, 180 and 240 minutes.
  Blood samples will be withdrawn from an intravenous cannula placed circa 10 minutes before the start of the study in the left antecubital vein. Samples will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C for the later measurement of PYY. All PYY assays will be performed using commercial radioimmunoassay kits at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.

SECONDARY OUTCOMES:
Changes in plasma concentrations of glucose and adiponectin over time as compared to baseline | During two study sessions lasting 4 hours each and performed at least two weeks apart. Blood samples will be taken twice at baseline and then hourly afterwards (between time-points 0 minutes and 240 minutes)
  Blood samples will be withdrawn from an intravenous cannula placed circa 10 minutes before the start of the study in the left antecubital vein. Glucose will be routinely measured in a certified laboratory (www.kimcl.at). Samples for the measurement of adiponectin will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C. All adiponectin assays will be performed using commercial kits at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.
Changes in plasma concentrations of cortisol, adrenaline and noradrenaline over time as compared to baseline | Timepoints -5, 0, 60, 120, 180 and 240 minutes.
  Blood samples will be withdrawn from an intravenous cannula placed circa 10 minutes before the start of the study in the left antecubital vein. Samples will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C for the later measurement of cortisol, adrenaline and noradrenaline. These assays will be performed using commercial kits used for routine purposes at a certified laboratory (www.kimcl.at) at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.
Changes in plasma concentrations of B-type natriuretic peptide (BNP) and atrial natriuretic peptide (ANP) over time as compared to baseline | Timepoints -5, 0, 60, 120, 180 and 240 minutes.
  Blood samples will be withdrawn from an intravenous cannula placed circa 10 minutes before the start of the study in the left antecubital vein in vacutainers containing heparin. Samples will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C for the later measurement of BNP and ANP. These assays will be performed using commercial kits used for routine purposes at a certified laboratory at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.
Changes in plasma concentrations of endothelial derived factors (endothelin, adrenomedullin and growth differentiation factor 15) over time as compared to baseline | Timepoints -5, 0, 60, 120, 180 and 240 minutes.
  Blood samples will be withdrawn from an intravenous cannula placed circa 10 minutes before the start of the study in the left antecubital vein. Samples will be immediately cooled on ice, centrifuged at 3000 rpm for 10 minutes and then stored at -20°C. All assays for adrenomedullin, endothelin and growth differentiation factor 15 will be performed using commercial kits used for routine purposes at a certified laboratory at the very end of the study with samples belonging to (both study days) one subject being measured within one kit.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Luger, MD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna
  - AKH, Medical University of Vienna, Vienna

REFERENCES:
- [Result] Vila G, Grimm G, Resl M, Heinisch B, Einwallner E, Esterbauer H, Dieplinger B, Mueller T, Luger A, Clodi M. B-type natriuretic peptide modulates ghrelin, hunger, and satiety in healthy men. Diabetes. 2012 Oct;61(10):2592-6. doi: 10.2337/db11-1466. Epub 2012 Jun 14. PMID 22698919